CLINICAL TRIAL: NCT05842512
Title: A Phase 2A, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Trial of ADI-PEG 20 or Placebo in Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Study of ADI-PEG 20 Versus Placebo in Subjects With NASH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POLARIS2023-001
Record Dates: First submitted 2023-01-20; First posted 2023-05-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: Nonalcoholic Steatohepatitis (NASH); Arginine; Arginine Deiminase; ADI-PEG 20; Pegargiminase
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — ADI PEG20

STUDY DESIGN:
Intervention Model Description: To evaluate efficacy and safety of ADI-PEG 20 or Placebo in patients with NASH
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a randomized, double-blind trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug: ADI-PEG 20 (Experimental): Dose: 36 mg/m2 given weekly Route of Administration: Intramuscular (IM)
  Interventions: Drug: ADI-PEG20
- Drug: Placebo (Placebo Comparator): Dose: 36 mg/m2 given weekly Route of Administration: Intramuscular (IM)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ADI-PEG20 — Treatment for NASH
  Other Names: Pegargiminase
  Arms: Drug: ADI-PEG 20
Other: Placebo — Treatment for NASH
  Arms: Drug: Placebo

SUMMARY:
Evaluate efficacy and safety of ADI-PEG 20 in patients with NASH

DETAILED DESCRIPTION:
The safety of ADI-PEG 20 will be assessed during the study through the reporting of adverse events (AEs), clinical laboratory tests, electrocardiogram (ECG), vital sign assessments, body weight, and concomitant medication usage.

An external Data Safety and Monitoring Committee (DSMB) that consists of two hepatologists and a statistician will review the safety of the study. The DSMB will convene after 10 subjects (approximately 5 per treatment group) have completed the Week 4 assessments. The DSMB will receive all reports of serious adverse events (SAEs) and convene as needed to monitor for safety.

The primary efficacy will be assessed via the absolute change from baseline in hepatic fat fraction measured by MRI-PDFF at Week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-lactating, pregnancy test negative females between 18 - 80 years of age with biopsy proven F1 - F4 (compensated cirrhosis, Child-Pugh A, score ≤6) NASH. Limit F1 fibrosis to ≤ 20% of total subject population.
2. Willingness to use appropriate contraceptive measures throughout study treatment and for 90 days thereafter (see Appendix A).
3. Body mass index (BMI) > 23 kg/m2
4. Must have confirmation of ≥ 5 % liver fat content on MRI-PDFF at screening.
5. Biopsy-proven NASH confirmed by a central pathologist. Must have had a liver biopsy either during the screening period or a historical biopsy conducted within the last 6 months prior to pre-screening with fibrosis stage 1 to 4 (F score, F1-F4) and a non-alcoholic fatty liver disease (NAFLD) activity score (NAS) of ≥ 4 with at least a score of 1 in each of the following NAS components:

   1. Steatosis (scored 0 to 3),
   2. Ballooning degeneration (scored 0 to 2), and
   3. Lobular inflammation (scored 0 to 3).
6. Must have no evidence of worsening of ALT and AST (within 50%) measurements within 2 months prior to screening (-8 weeks) visits.
7. Screening laboratory parameters, as determined by the central laboratory:

   1. Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min, as calculated by the Cockcroft- Gault equation;
   2. HbA1c ≤ 9.5% (or serum fructosamine ≤ 381 μmol if HbA1c is unable to be resulted);
   3. Hemoglobin ≥ 11 g/dL;
   4. INR ≤ 1.3, unless due to therapeutic anticoagulation;
   5. Direct bilirubin ≤ 0.5 mg/dL;
   6. Total bilirubin ≤ 1.3 x upper limit of normal (ULN), unless due to an alternate etiology such as Gilbert's syndrome or hemolytic anemia;
   7. Creatinine kinase < 3 x ULN;
   8. Platelet count ≥ 150,000/μL;
   9. Serum triglyceride level ≤ 500 mg/dL;
   10. ALT < 6 x ULN;
   11. AST < 6 x ULN;
   12. ALP < 2 x ULN.
8. FibroScan® measurement > 7.0 kPa and < 20.0 kPa.
9. Subjects on non-insulin dependent diabetic, weight loss, or lipid-modifying medication(s) must be on stable dose(s) for at least 3 months prior to the diagnostic liver biopsy through randomization.
10. Subjects on vitamin E and pioglitazone must maintain a stable dosage before the diagnostic liver biopsy and during the study period.

Exclusion Criteria:

1. Weight gain or loss > 5% in the 3 months prior to randomization or > 10% in the 6 months prior to screening.
2. Type 1 and insulin-dependent Type 2 diabetes.
3. Poorly controlled hypertension (blood pressure [BP] > 160/100 mmHg).
4. Prior history of decompensated liver disease including ascites, hepatic encephalopathy (HE), or variceal bleeding.
5. Chronic hepatitis B virus (HBV) infection (hepatitis B surface antigen [HBsAg] positive.
6. Chronic hepatitis C virus (HCV) infection (HCV antibody [Ab] and HCV ribonucleic acid [RNA] positive). Subjects cured of HCV infection less than 1 year prior (based on date of RNA polymerase chain reaction [PCR] negative confirmation following conclusion of treatment) to the screening visit are not eligible.
7. Prior or planned (during the study period) bariatric surgery (e.g., gastroplasty, roux-en-Y gastric bypass), surgery reversal or removal of intragastric balloon > 2 years prior to enrollment would be eligible.
8. Other causes of liver disease based on medical history and/or centralized review of liver histology, including but not limited to alcoholic liver disease, autoimmune disorders (e.g., primary biliary cholangitis [PBC], primary sclerosing cholangitis [PSC], autoimmune hepatitis), drug-induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1-antitrypsin deficiency requiring treatment.
9. History of liver transplantation.
10. Subjects with primary cancer, including co-existent second malignancy, with the exception of primary solid tumor with no known active disease present in the opinion of the Investigator which will not affect subject outcome in the setting of current diagnosis.
11. Alcohol intake above an average limit of 2 drinks per day for women and 3 drinks per day for men. An alcoholic drink is defined as 12 ounces of regular beer, which is usually about 5% alcohol, 5 ounces of wine, which is typically about 12% alcohol, and 1.5 ounces of distilled spirits, which is about 40% alcohol.
12. Human immunodeficiency virus (HIV) infection.
13. Unstable cardiovascular disease in the 6 months prior to screening.
14. Life expectancy less than 2 years.
15. Use of any investigational medication within 30 days or within 5 half-lives of the investigational medication, whichever is longer, prior to screening and throughout the study is prohibited.
16. Subjects with a history of (12 months prior to baseline) or current use of prescription drugs associated with liver steatosis (e.g., methotrexate, amiodarone, high-dose estrogen, tamoxifen, systemic steroids, anabolic steroids, valproic acid) should be excluded. However, subjects currently using silymarin should maintain their current dosage throughout the trial period.
17. Contraindication of magnetic resonance imaging. These include but are not limited to devices or metal foreign bodies, such as Pacemaker, defibrillator or wires other than sternal wires, metallic foreign body in the eye, "triggerfish" contact lens, gastric reflux device, and insulin pumps.
18. MELD score >12
19. Subjects with esophageal or gastric varices with recent bleeding episodes (within 1 year).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Determine Efficacy of ADI-PEG 20 vs Placebo in the treatment of fatty liver as assessed by change in hepatic fat fraction | 24 Weeks
  Evaluate absolute change from baseline in hepatic fat fraction assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF) at Week 24

SECONDARY OUTCOMES:
Assess the Efficacy of ADI-PEG 20 vs Placebo reflected in the percent change from baseline in hepatic fat fraction at week 24 | 24 Weeks
  Evaluate percent change from baseline in hepatic fat fraction assessed by MRI-PDFF at Week 24
Assess the safety of ADI-PEG 20 in subjects with NASH | 24 Weeks
  Evaluate the change from baseline in ALT at Weeks 12 and 24.
Assess the safety and tolerability of ADI-PEG 20 in subjects with NASH | 24 Weeks
  Laboratory tests and clinical adverse events

CONTACTS AND LOCATIONS:
Overall Officials: John S Bomalaski, Study Director — Polaris Group
Locations (10):
- Taiwan (10):
  - Ditmanson Medical Foundation Chiayi Christian Hospital；Chiayi Christian Hospital (CYCH), Chiayi City, Taiwan
  - Kaohsiung Medical University Chung-Ho Memorial Hospital(KMUH), Kaohsiung, Taiwan
  - E-Da Hospital (EDH), Kaohsiung, Taiwan
  - Chang Gung Medical Foundation-Kaohsiung (CGMF-KS), Kaohsiung, Taiwan
  - Chang Gung Medical Foundation-Keelung (CGMF-KL), Keelung, Taiwan
  - National Cheng Kung University Hospital (NCKUH), Tainan, Taiwan
  - National Taiwan University Hospital (NTUH), Taipei, Taiwan
  - Taipei Veterans General Hospital (TPVGH), Taipei, Taiwan
  - Fu Jen Catholic University Hospital (FJCUH), Taipei, Taiwan
  - Chang Gung Medical Foundation-Linkou (CGMF-LK), Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No